CLINICAL TRIAL: NCT00740038
Title: Study of Stress Management and Exercise Intervention During Cancer Chemotherapy
Brief Title: Support for People Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-13782; ACS RSGPB-05-0243-01 (CPPB)
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2011-08

CONDITIONS: Quality of Life; Cancer
Keywords: Stress Management; Quality of Life; Exercise; Cancer; Chemotherapy
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Coping Skills; Autogenic Training; Imagery, Psychotherapy; Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Active Control: Usual Care
  Interventions: Behavioral: Usual care
- 2 (Experimental): Stress Management Intervention
  Interventions: Behavioral: Stress Management training
- 3 (Experimental): Exercise Intervention
  Interventions: Behavioral: Exercise Training
- 4 (Experimental): Combined Stress Management and Exercise Intervention
  Interventions: Behavioral: Combined stress management and exercise training

INTERVENTIONS:
Behavioral: Stress Management training — Self-administered stress management training comprising 10 minute introduction by staff, & provision of DVD, CD,brochure, and workbook. Materials provide overview of sources of stress during chemotherapy, and instruction in cognitive-behavioral stress management techniques (paced abdominal breathing, progressive muscle relaxation with guided imagery, and use of coping self-statements). Daily use is encouraged over 13-14 weeks of the study.
  Other Names: Coping techniques; Cognitive-behavioral; stress management; Progressive muscle relaxation; Deep Breathing; Guided Imagery; Positive self-statements coping
  Arms: 2
Behavioral: Exercise Training — Home-based exercise (walking) program: brief introduction by staff (10 minutes) and provision of packet with DVD, brochure, workbook, pedometer (electronic step counter) along with instructions on initiating and maintaining a walking program. Dose Recommendations: 3-5 exercise session per week for at least 20-30 minutes at maximum intensity of 50 to 75% of their estimated heart rate reserve (RPE of 11-13) which is calculated based on their age and resting pulse.
  Other Names: Exercise program; Walking program; home-based exercise; exercise during chemotherapy
  Arms: 3
Behavioral: Usual care — Usual psychosocial care and provision of NCI booklet, Chemotherapy and You (NCI, 1999) which gives general feedback about fitness testing, exercise and stress management during chemotherapy. Recommended to read booklet at least once.
  Other Names: Active control group; Information on chemotherapy
  Arms: 1
Behavioral: Combined stress management and exercise training — Home-based, self-administered stress management and exercise (walking) program: brief introduction by staff and provision of DVD, CD, brochure, pedometer, workbook. Dose Recommendations: walking/exercise program (3-5 times per week for at least 20-30 minutes) and use of CD (progressive muscle relaxation with guided imagery) and coping statements once per day.
  Other Names: Stress management and exercise; Exercise and stress management; exercise during chemotherapy; Progressive muscle relaxation; Guided Imagery; Coping self-statements; walking program
  Arms: 4

SUMMARY:
Chemotherapy adversely affects quality of life in cancer patients. Both stress management training and exercise training have been shown to improve quality of life. These two types of training have not been directly compared for chemotherapy patients.

This study seeks to evaluate the separate and combined effects of stress management training and exercise training on quality of life during chemotherapy treatment. Participants receive either a home-based, self-administered program in 1 of 3 types (stress management, exercise, or stress management + exercise) or usual care (reading materials). It is hypothesized that the combined program (stress management + exercise) will be significantly associated with better quality of life than the usual care group, the exercise only group, and the stress management only group. All participants are assessed at 3 timepoints: before they begin chemotherapy, 6 weeks after their first chemotherapy infusion, and 12 weeks after their first infusion.

ELIGIBILITY:
Inclusion Criteria: participants must:

* Be diagnosed with cancer
* Be scheduled to receive cytotoxic chemotherapy for at least 14 weeks
* Be ≥18 years of age or older
* Have an ECOG performance status of 0, 1, or 2
* Be capable of speaking and reading English
* Be able to provide informed consent

Exclusion Criteria:

* ECOG of 3 or greater
* Presence of contraindications to participating in moderate intensity exercise including:

  1. . metastases to weight-bearing sites (spine, pelvis, lower extremities)
  2. . active infections
  3. . cardiomyopathy or congestive heart failure
  4. . severe pulmonary or ventilatory disease (FEV 1.0<50%)
  5. . large pleural effusions or pericardial effusions
  6. . anemia (Hgb <8g/dL)
  7. . neutropenia (absolute neutrophil count < 0.05 x 10(9th)/L)
  8. . severe osteoporosis (> 2.5 SD below age and gender norms)
  9. . thrombocytopenia (platelets < 20 x 10(9th)/L)
  10. . hyponatremia (Na+ < 130 mmol/L)
  11. . hypokalemia (K+ ≤ 3.0 mmol/L)
  12. . hypercalcemia (Ca++ > 6.5 mmol/L)
  13. . abnormal ECG
  14. . sensorimotor deficits sufficient to impede unassisted walking
* Receipt of intravenous chemotherapy administration in the past 2 months
* Prescription for chronotropic, sympathomimetic, or inotropic/vasoactive medications
* Presence of other contraindications as determined by the attending oncologist and research staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2006-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Survey-Short Form (SF-36, acute) | pre-chemotherapy baseline, 6 weeks post-1st infusion, & 12-weeks post-initial infusion

SECONDARY OUTCOMES:
Center for Epidemiological Studies-Depression (CES-D) | pre-chemotherapy baseline, 6- & 12- weeks post-baseline
Beck Anxiety Inventory (BAI) | pre-chemotherapy baseline, 6- & 12-weeks post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Jacobsen, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Background] Courneya KS, Mackey JR, & Quinney HA. Neoplasms. In Myers, Herbert, Humphrey (eds): American College of Sports Medicine resources for clinical exercise physiology: musculoskeletal, neuromuscular, immunologic, and hematologic conditions. New York: Lippincott.
- [Background] Courneya KS, Mackey JR, Bell GJ, Jones LW, Field CJ, Fairey AS. Randomized controlled trial of exercise training in postmenopausal breast cancer survivors: cardiopulmonary and quality of life outcomes. J Clin Oncol. 2003 May 1;21(9):1660-8. doi: 10.1200/JCO.2003.04.093. PMID 12721239
- [Background] Courneya KS, Friedenreich CM, Sela RA, Quinney HA, Rhodes RE, Handman M. The group psychotherapy and home-based physical exercise (group-hope) trial in cancer survivors: physical fitness and quality of life outcomes. Psychooncology. 2003 Jun;12(4):357-74. doi: 10.1002/pon.658. PMID 12748973
- [Background] Jacobsen PB, Meade CD, Stein KD, Chirikos TN, Small BJ, Ruckdeschel JC. Efficacy and costs of two forms of stress management training for cancer patients undergoing chemotherapy. J Clin Oncol. 2002 Jun 15;20(12):2851-62. doi: 10.1200/JCO.2002.08.301. PMID 12065562
- [Derived] Phillips KM, Jim HS, Small BJ, Tanvetyanon T, Roberts WS, Jacobsen PB. Effects of self-directed stress management training and home-based exercise on stress management skills in cancer patients receiving chemotherapy. Stress Health. 2012 Dec;28(5):368-75. doi: 10.1002/smi.2450. Epub 2012 Sep 13. PMID 22972771